CLINICAL TRIAL: NCT05746390
Title: Home Alone: Developing a Home-Based Intervention for People With Cognitive Impairment Who Live Alone
Brief Title: Home Alone: An Intervention for People With Cognitive Impairment Who Live Alone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00017313
Record Dates: First submitted 2023-02-10; First posted 2023-02-27 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Cognitive Impairment; Dementia; Memory Loss
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Memory Disorders | interventions — Home Environment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home Alone Intervention (Experimental): Home Alone is a semi-structured intervention, tailored to address the individual needs and concerns of the older adult. The participant will engage in about seven psychoeducational coaching sessions, each lasting approximately one hour.
  The intervention has two key foci:
  1. increasing or maintaining home safety and comfort
  2. increasing scheduled social engagements and activities.
  Sessions are also designed to identify formal and informal services and supports to improve to increase assistance and ability to live independently for as long as safely possible. The sessions take place either in-person or remotely (via secure video conferencing or telephone). Ad hoc/ongoing sessions may be provided as needed.
  Interventions: Behavioral: Home Alone

INTERVENTIONS:
Behavioral: Home Alone — See Home Alone description.

SUMMARY:
The goal of this clinical trial is to evaluate a program for adults who live alone and have some cognitive impairment (CI) to see if it is useful and acceptable. This program aims to help older adults with cognitive impairment who live alone to be engaged and active, as well as safe at home. The investigators want to see how useful this program is and how it can be improved.

The specific aims are:

* Specific Aim 1: Develop and Adapt Home Alone to Prepare for Pilot Testing.
* Specific Aim 2: Pilot Test a Revised Version of Home Alone.

Phase I participants will be asked to:

* Participate for 3 months
* Complete 3 surveys
* Complete 7 1-hour meetings on a weekly basis with a coach
* Complete a final interview

Phase II participants will be asked to:

* Participate for 6 months
* Complete 3 surveys
* Complete 7 1-hour meetings on a weekly basis with a coach
* A sub-sample will be asked to complete a final interview

DETAILED DESCRIPTION:
The primary goal of this proposal is to establish the feasibility, acceptability, and appropriateness of a novel intervention, "Home Alone." Home Alone will be targeted to older persons with CI or Mild Cognitive Impairment (MCI) who live alone in the community. This National Institute on Aging (NIA) Stage I effort will adapt and tailor established, evidence-based mental health and dementia care intervention models (behavioral activation, Skills2Care®, Tailored Activity Program) to reduce environmental stress and enhance engagement in desired activities to improve social well-being and maintain cognition and function for those who live alone with CI. Relying on a robust, mixed methods strategy and an implementation science lens at the outset of intervention development, the investigators seek to position Home Alone as a scalable program that, as its efficacy and effectiveness is determined in subsequent trials, is primed for widespread dissemination and adoption in home-based and community contexts.

The Specific Aims are as follows:

Specific Aim 1 (Phase I): Develop and Adapt Home Alone to Prepare for Pilot Testing. The investigators will identify treatment components and examine feasibility and relevance by obtaining insights from 15 persons with CI who live alone and participate in the Home Alone intervention over a 3-month period. The investigators will utilize the Phase I period to determine whether various elements of Home Alone (e.g., delivery mode, length, and other intervention characteristics) require adaptation. The investigators will use a convergent parallel mixed methods design (i.e., the collection and analysis of quantitative and qualitative data concurrently) when doing so. Through analysis of the various quantitative and qualitative data elements to inform adaptation, the investigators will finalize and refine Home Alone prior to project Phase II (Specific Aim 2).

Specific Aim 2 (Phase II): Pilot Test a Revised Version of Home Alone. This R21 project will evaluate the following indices of implementation potential over a 6-month period: whether Home Alone is carried out as intended and is feasible (the degree to which Home Alone can be successfully delivered); acceptable (Home Alone is agreeable and satisfactory among users), and useful (participants perceive benefit from the Home Alone intervention). A sequential explanatory mixed methods design (a quantitative component followed by a qualitative component) will be utilized to pilot test Home Alone. The investigators will enroll 50 persons living alone with CI over a 6-month period. The investigators will also examine whether key empirical outcomes (perceived loneliness; activity engagement; measures of cognition and functional dependence) change over a 6-month period. Available qualitative data will provide information on how and why Home Alone was beneficial or not for persons with CI and allow for greater understanding of the intervention's mechanisms of benefit.

Home Alone combines Behavioral Activation (BA) with other evidence-based intervention approaches (i.e., Tailored Activity Program (TAP); Skills2Care®) that target the environment in order to tailor activity that is fulfilling and meaningful to persons with CI. An additional intervention component that will be incorporated in Home Alone includes environmental assessments that help the person with CI by removing objects and improving lighting and safety in areas of the home where a desired and meaningful activity will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* 55 years of age or older
* Lives alone in a non-residential setting
* Either 1) provider diagnosis of MCI, 2) Montreal Cognitive Assessment by telephone (T-MoCA) score between 13 and 18, and/or 3) subjective endorsement of memory impairment on screening
* Resides in the US
* Demonstrates capacity to consent

Exclusion Criteria:

Those who do not meet the inclusion criteria above are not eligible. Additionally, researchers would exclude those who:

* Live in assisted living, a group care home, or similar residential setting that provides care and services
* Are not English speaking
* Are currently participating in any other type of service that provides one-to-one psychosocial consultation or independent living coaching
* Have a new or worsening mental health condition and are not receiving ongoing treatment
* Have not remained on a stable psychotropic medications dosage, such as antidepressants, anxiolytics, or anti-psychotics, for the prior three months
* Are not willing/interested in participating or cannot actively participate in the intervention, per researcher discretion

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
Acceptability of Intervention | Phase I at 1 month
  Acceptability of Intervention Measure - 4 item scale evaluating program acceptability. The measure evaluates the likeability of the intervention (e.g. I like the intervention; I welcome the intervention; the intervention meets my approval; the intervention is appealing to me). Items are rated on a scale of agreement (completely disagree, disagree, neither agree or disagree, agree, completely agree). Scores range from 4-20, with higher scores indicating higher levels of acceptability.
Acceptability of Intervention | Phase I at 3 months
  Acceptability of Intervention Measure - 4 item scale evaluating program acceptability. The measure evaluates the likeability of the intervention (e.g. I like the intervention; I welcome the intervention; the intervention meets my approval; the intervention is appealing to me). Items are rated on a scale of agreement (completely disagree, disagree, neither agree or disagree, agree, completely agree). Scores range from 4-20, with higher scores indicating higher levels of acceptability.
Acceptability of Intervention | Phase II at 3 months
  Acceptability of Intervention Measure - 4 item scale evaluating program acceptability. The measure evaluates the likeability of the intervention (e.g. I like the intervention; I welcome the intervention; the intervention meets my approval; the intervention is appealing to me). Items are rated on a scale of agreement (completely disagree, disagree, neither agree or disagree, agree, completely agree). Scores range from 4-20, with higher scores indicating higher levels of acceptability.
Acceptability of Intervention | Phase II at 6 months
  Acceptability of Intervention Measure - 4 item scale evaluating program acceptability. The measure evaluates the likeability of the intervention (e.g. I like the intervention; I welcome the intervention; the intervention meets my approval; the intervention is appealing to me). Items are rated on a scale of agreement (completely disagree, disagree, neither agree or disagree, agree, completely agree). Scores range from 4-20, with higher scores indicating higher levels of acceptability.
Feasibility of Intervention | Phase I at 1 month
  Feasibility of Intervention Measure - 4 item scale evaluating program feasibility; The measure includes four statements about the feasibility of intervention implementation (ex. the intervention seems implementable; the intervention seems doable; the intervention seems possible; the intervention seems easy to use). Items are rated on a five-point scale (completely disagree, disagree, neither agree or disagree, agree, completely agree). Scores range from 4-20. Higher scores indicate greater feasibility.
Feasibility of Intervention | Phase I at 3 months
  Feasibility of Intervention Measure - 4 item scale evaluating program feasibility; The measure includes four statements about the feasibility of intervention implementation (ex. the intervention seems implementable; the intervention seems doable; the intervention seems possible; the intervention seems easy to use). Items are rated on a five-point scale (completely disagree, disagree, neither agree or disagree, agree, completely agree). Scores range from 4-20. Higher scores indicate greater feasibility.
Feasibility of Intervention | Phase II at 3 months
  Feasibility of Intervention Measure - 4 item scale evaluating program feasibility; The measure includes four statements about the feasibility of intervention implementation (ex. the intervention seems implementable; the intervention seems doable; the intervention seems possible; the intervention seems easy to use). Items are rated on a five-point scale (completely disagree, disagree, neither agree or disagree, agree, completely agree). Scores range from 4-20. Higher scores indicate greater feasibility.
Feasibility of Intervention | Phase II at 6 months
  Feasibility of Intervention Measure - 4 item scale evaluating program feasibility; The measure includes four statements about the feasibility of intervention implementation (ex. the intervention seems implementable; the intervention seems doable; the intervention seems possible; the intervention seems easy to use). Items are rated on a five-point scale (completely disagree, disagree, neither agree or disagree, agree, completely agree). Scores range from 4-20. Higher scores indicate greater feasibility.
Intervention Appropriateness | Phase I at 1 month
  Intervention Appropriateness Measure - 4 item scale evaluating program appropriateness; The measure includes four statements about the feasibility of intervention implementation (ex. the intervention seems fitting; the intervention seems suitable; the intervention seems applicable; the intervention seems liked a good match). Items are rated on a five-point scale (completely disagree, disagree, neither agree or disagree, agree, completely agree). Scores range from 4-20. Higher scores indicate greater appropriateness.
Intervention Appropriateness | Phase I at 3 months
  Intervention Appropriateness Measure - 4 item scale evaluating program appropriateness; The measure includes four statements about the feasibility of intervention implementation (ex. the intervention seems fitting; the intervention seems suitable; the intervention seems applicable; the intervention seems liked a good match). Items are rated on a five-point scale (completely disagree, disagree, neither agree or disagree, agree, completely agree). Scores range from 4-20. Higher scores indicate greater appropriateness.
Intervention Appropriateness | Phase II at 3 months
  Intervention Appropriateness Measure - 4 item scale evaluating program appropriateness; The measure includes four statements about the feasibility of intervention implementation (ex. the intervention seems fitting; the intervention seems suitable; the intervention seems applicable; the intervention seems liked a good match). Items are rated on a five-point scale (completely disagree, disagree, neither agree or disagree, agree, completely agree). Scores range from 4-20. Higher scores indicate greater appropriateness.
Intervention Appropriateness | Phase II at 6 months
  Intervention Appropriateness Measure - 4 item scale evaluating program appropriateness; The measure includes four statements about the feasibility of intervention implementation (ex. the intervention seems fitting; the intervention seems suitable; the intervention seems applicable; the intervention seems liked a good match). Items are rated on a five-point scale (completely disagree, disagree, neither agree or disagree, agree, completely agree). Scores range from 4-20. Higher scores indicate greater appropriateness.
Intervention Treatment Receipt | Phase I at 1 month
  Intervention Treatment Receipt Checklist Measure - Eleven item checklist designed for study, measuring whether the coach delivered key aspects of the intervention. The measure includes 10 Likert scale items and one open-ended question on the appropriateness and acceptability of Home Alone and the extent to which Home Alone helps participants with CI modify their environment, engage in pleasant activities, and access social and other resources. The 10 items are scored on a 5 point Likert scale with a total score ranging from 0-50, where higher scores indicate greater treatment fidelity and acceptability of the intervention.
Intervention Treatment Receipt | Phase I at 3 months
  Intervention Treatment Receipt Checklist Measure - Eleven item checklist designed for study, measuring whether the coach delivered key aspects of the intervention. The measure includes 10 Likert scale items and one open-ended question on the appropriateness and acceptability of Home Alone and the extent to which Home Alone helps participants with CI modify their environment, engage in pleasant activities, and access social and other resources. The 10 items are scored on a 5 point Likert scale with a total score ranging from 0-50, where higher scores indicate greater treatment fidelity and acceptability of the intervention.
Intervention Treatment Receipt | Phase II at 3 months
  Intervention Treatment Receipt Checklist Measure - Eleven item checklist designed for study, measuring whether the coach delivered key aspects of the intervention. The measure includes 10 Likert scale items and one open-ended question on the appropriateness and acceptability of Home Alone and the extent to which Home Alone helps participants with CI modify their environment, engage in pleasant activities, and access social and other resources. The 10 items are scored on a 5 point Likert scale with a total score ranging from 0-50, where higher scores indicate greater treatment fidelity and acceptability of the intervention.
Intervention Treatment Receipt | Phase II at 6 months
  Intervention Treatment Receipt Checklist Measure - Eleven item checklist designed for study, measuring whether the coach delivered key aspects of the intervention. The measure includes 10 Likert scale items and one open-ended question on the appropriateness and acceptability of Home Alone and the extent to which Home Alone helps participants with CI modify their environment, engage in pleasant activities, and access social and other resources. The 10 items are scored on a 5 point Likert scale with a total score ranging from 0-50, where higher scores indicate greater treatment fidelity and acceptability of the intervention.

SECONDARY OUTCOMES:
Social Well-being/Loneliness (Social contact and Support) | Phase I at baseline
  Lubben Social Network Scale-6 6 item scale evaluating social engagement; Items assess social contact and support including family and friends; Scores range from 0 to 30, with higher scores representing more social engagement.
Social Well-being/Loneliness (Social contact and Support) | Phase I at 1 month
  Lubben Social Network Scale-6 6 item scale evaluating social engagement; Items assess social contact and support including family and friends; Scores range from 0 to 30, with higher scores representing more social engagement.
Social Well-being/Loneliness (Social contact and Support) | Phase I at 3 months
  Lubben Social Network Scale-6 6 item scale evaluating social engagement; Items assess social contact and support including family and friends; Scores range from 0 to 30, with higher scores representing more social engagement.
Social Well-being/Loneliness (Social contact and Support) | Phase II at baseline
  Lubben Social Network Scale-6 6 item scale evaluating social engagement; Items assess social contact and support including family and friends; Scores range from 0 to 30, with higher scores representing more social engagement.
Social Well-being/Loneliness (Social contact and Support) | Phase II at 3 months
  Lubben Social Network Scale-6 6 item scale evaluating social engagement; Items assess social contact and support including family and friends; Scores range from 0 to 30, with higher scores representing more social engagement.
Social Well-being/Loneliness (Social contact and Support) | Phase II at 6 months
  Lubben Social Network Scale-6 6 item scale evaluating social engagement; Items assess social contact and support including family and friends; Scores range from 0 to 30, with higher scores representing more social engagement.
Social Well-being/Loneliness (Loneliness) | Phase I at baseline
  De Jong Gierveld Loneliness Scale (Short - 6 items) will measure emotional and social loneliness; Scores range from 1-6. Higher scores indicate greater levels of loneliness.
Social Well-being/Loneliness (Loneliness) | Phase I at 1 month
  De Jong Gierveld Loneliness Scale (Short - 6 items) will measure emotional and social loneliness; Scores range from 1-6. Higher scores indicate greater levels of loneliness.
Social Well-being/Loneliness (Loneliness) | Phase I at 3 months
  De Jong Gierveld Loneliness Scale (Short - 6 items) will measure emotional and social loneliness; Scores range from 1-6. Higher scores indicate greater levels of loneliness.
Social Well-being/Loneliness (Loneliness) | Phase II at baseline
  De Jong Gierveld Loneliness Scale (Short - 6 items) will measure emotional and social loneliness; Scores range from 1-6. Higher scores indicate greater levels of loneliness.
Social Well-being/Loneliness (Loneliness) | Phase II at 3 months
  De Jong Gierveld Loneliness Scale (Short - 6 items) will measure emotional and social loneliness; Scores range from 1-6. Higher scores indicate greater levels of loneliness.
Social Well-being/Loneliness (Loneliness) | Phase II at 6 months
  De Jong Gierveld Loneliness Scale (Short - 6 items) will measure emotional and social loneliness; Scores range from 1-6. Higher scores indicate greater levels of loneliness.
Social Well-being/Loneliness (Well-being) | Phase I at baseline
  Geriatric Depression Scale-Short Form -15 items measuring emotional well-being; scores range from 0-15; Scores under 5 indicate that depression is unlikely, scores of 5 or more suggest depression.
Social Well-being/Loneliness (Well-being) | Phase I at 1 month
  Geriatric Depression Scale-Short Form -15 items measuring emotional well-being; scores range from 0-15; Scores under 5 indicate that depression is unlikely, scores of 5 or more suggest depression.
Social Well-being/Loneliness (Well-being) | Phase I at 3 months
  Geriatric Depression Scale-Short Form -15 items measuring emotional well-being; scores range from 0-15; Scores under 5 indicate that depression is unlikely, scores of 5 or more suggest depression.
Social Well-being/Loneliness (Well-being) | Phase II at baseline
  Geriatric Depression Scale-Short Form -15 items measuring emotional well-being; scores range from 0-15; Scores under 5 indicate that depression is unlikely, scores of 5 or more suggest depression.
Social Well-being/Loneliness (Well-being) | Phase II at 3 months
  Geriatric Depression Scale-Short Form -15 items measuring emotional well-being; scores range from 0-15; Scores under 5 indicate that depression is unlikely, scores of 5 or more suggest depression.
Social Well-being/Loneliness (Well-being) | Phase II at 6 months
  Geriatric Depression Scale-Short Form -15 items measuring emotional well-being; scores range from 0-15; Scores under 5 indicate that depression is unlikely, scores of 5 or more suggest depression.
Activity/Engagement | Phase I at baseline
  Pleasant Events Schedule: Alzheimer's Disease (AD) short form - 20 activity items measured on a scale divided into two parts. The first part of the scale measures frequency of participation and availability of the event (ltems are rated from 0 to 2; total scores can range from 0 to 40). The second part of the scale assesses current and/or past enjoyment of those activities (ltems are rated from 0 to 1; total scores can range from 0 to 20). Higher scores indicate higher levels of activity on both subscales.
Activity/Engagement | Phase I at 1 month
  Pleasant Events Schedule: Alzheimer's Disease (AD) short form - 20 activity items measured on a scale divided into two parts. The first part of the scale measures frequency of participation and availability of the event (ltems are rated from 0 to 2; total scores can range from 0 to 40). The second part of the scale assesses current and/or past enjoyment of those activities (ltems are rated from 0 to 1; total scores can range from 0 to 20). Higher scores indicate higher levels of activity on both subscales.
Activity/Engagement | Phase I at 3 months
  Pleasant Events Schedule: Alzheimer's Disease (AD) short form - 20 activity items measured on a scale divided into two parts. The first part of the scale measures frequency of participation and availability of the event (ltems are rated from 0 to 2; total scores can range from 0 to 40). The second part of the scale assesses current and/or past enjoyment of those activities (ltems are rated from 0 to 1; total scores can range from 0 to 20). Higher scores indicate higher levels of activity on both subscales.
Activity/Engagement | Phase II at baseline
  Pleasant Events Schedule: Alzheimer's Disease (AD) short form - 20 activity items measured on a scale divided into two parts. The first part of the scale measures frequency of participation and availability of the event (ltems are rated from 0 to 2; total scores can range from 0 to 40). The second part of the scale assesses current and/or past enjoyment of those activities (ltems are rated from 0 to 1; total scores can range from 0 to 20). Higher scores indicate higher levels of activity on both subscales.
Activity/Engagement | Phase II at 3 months
  Pleasant Events Schedule: Alzheimer's Disease (AD) short form - 20 activity items measured on a scale divided into two parts. The first part of the scale measures frequency of participation and availability of the event (ltems are rated from 0 to 2; total scores can range from 0 to 40). The second part of the scale assesses current and/or past enjoyment of those activities (ltems are rated from 0 to 1; total scores can range from 0 to 20). Higher scores indicate higher levels of activity on both subscales.
Activity/Engagement | Phase II at 6 months
  Pleasant Events Schedule: Alzheimer's Disease (AD) short form - 20 activity items measured on a scale divided into two parts. The first part of the scale measures frequency of participation and availability of the event (ltems are rated from 0 to 2; total scores can range from 0 to 40). The second part of the scale assesses current and/or past enjoyment of those activities (ltems are rated from 0 to 1; total scores can range from 0 to 20). Higher scores indicate higher levels of activity on both subscales.
Cognition | Phase I at screening
  Telephone Montreal Cognitive Assessment (T-MoCA) - measure assessing 8 areas of cognition used over the phone to screen for Mild Cognitive Impairment; scores range from 0-22; with higher scores indicating better cognitive functioning. Scores 18 or below suggest mild cognitive dysfunction.
Cognition | Phase I at 1 month
  Telephone Montreal Cognitive Assessment (T-MoCA) - measure assessing 8 areas of cognition used over the phone to screen for Mild Cognitive Impairment; scores range from 0-22; with higher scores indicating better cognitive functioning. Scores 18 or below suggest cognitive dysfunction.
Cognition | Phase I at 3 months
  Telephone Montreal Cognitive Assessment (T-MoCA) - measure assessing 8 areas of cognition used over the phone to screen for Mild Cognitive Impairment; scores range from 0-22; with higher scores indicating better cognitive functioning. Scores 18 or below suggest mild cognitive dysfunction.
Cognition | Phase II at screening
  Telephone Montreal Cognitive Assessment (T-MoCA) - measure assessing 8 areas of cognition used over the phone to screen for Mild Cognitive Impairment; scores range from 0-22; with higher scores indicating better cognitive functioning. Scores 18 or below suggest mild cognitive dysfunction.
Cognition | Phase II at 3 months
  Telephone Montreal Cognitive Assessment (T-MoCA) - measure assessing 8 areas of cognition used over the phone to screen for Mild Cognitive Impairment; scores range from 0-22; with higher scores indicating better cognitive functioning. Scores 18 or below suggest mild cognitive dysfunction.
Cognition | Phase II at 6 months
  Telephone Montreal Cognitive Assessment (T-MoCA) - measure assessing 8 areas of cognition used over the phone to screen for Mild Cognitive Impairment; scores range from 0-22; with higher scores indicating better cognitive functioning. Scores 18 or below suggest mild cognitive dysfunction.
Functional Dependence - Activities of Daily Living (ADL)/Independent Activities of Daily Living (IADL) | Phase I at baseline
  Fifteen item scale created from Katz Activities of Daily Living- 6 item scale measuring ability to perform activities of daily living, 8 items from the Lawton Independent Activities of Daily Living scale assessing 8 domains of independent living skills (including shopping and taking medications) and 1 item on hygiene from the Routine Task Inventory; Scores range from 0-30 with higher scores needing more help with ADL/IADLs.
Functional Dependence - Activities of Daily Living (ADL)/Independent Activities of Daily Living (IADL) | Phase I at 1 month
  Fifteen item scale created from Katz Activities of Daily Living- 6 item scale measuring ability to perform activities of daily living, 8 items from the Lawton Independent Activities of Daily Living scale assessing 8 domains of independent living skills (including shopping and taking medications) and 1 item on hygiene from the Routine Task Inventory; Scores range from 0-30 with higher scores needing more help with ADL/IADLs.
Functional Dependence - Activities of Daily Living (ADL)/Independent Activities of Daily Living (IADL) | Phase I at 3 months
  Fifteen item scale created from Katz Activities of Daily Living- 6 item scale measuring ability to perform activities of daily living, 8 items from the Lawton Independent Activities of Daily Living scale assessing 8 domains of independent living skills (including shopping and taking medications) and 1 item on hygiene from the Routine Task Inventory; Scores range from 0-30 with higher scores needing more help with ADL/IADLs.
Functional Dependence - Activities of Daily Living (ADL)/Independent Activities of Daily Living | Phase II at baseline
  Fifteen item scale created from Katz Activities of Daily Living- 6 item scale measuring ability to perform activities of daily living, 8 items from the Lawton Independent Activities of Daily Living scale assessing 8 domains of independent living skills (including shopping and taking medications) and 1 item on hygiene from the Routine Task Inventory; Scores range from 0-30 with higher scores needing more help with ADL/IADLs.
Functional Dependence - Activities of Daily Living (ADL)/Independent Activities of Daily Living | Phase II at 3 months
  Fifteen item scale created from Katz Activities of Daily Living- 6 item scale measuring ability to perform activities of daily living, 8 items from the Lawton Independent Activities of Daily Living scale assessing 8 domains of independent living skills (including shopping and taking medications) and 1 item on hygiene from the Routine Task Inventory; Scores range from 0-30 with higher scores needing more help with ADL/IADLs.
Functional Dependence - Activities of Daily Living (ADL)/Independent Activities of Daily Living (IADL) | Phase II at 6 months
  Fifteen item scale created from Katz Activities of Daily Living- 6 item scale measuring ability to perform activities of daily living, 8 items from the Lawton Independent Activities of Daily Living scale assessing 8 domains of independent living skills (including shopping and taking medications) and 1 item on hygiene from the Routine Task Inventory; Scores range from 0-30 with higher scores needing more help with ADL/IADLs.
Functional Dependence (Physical functioning) | Phase I at baseline.
  US Health Interview Survey - assesses engagement in physical activities in the prior two weeks. A composite index of physical activity is computed by summing the products of the number of minutes in each activity (9 are listed and there is an open response "other" option) and how many times in the past two weeks the engaged in the activity for the 9 activities and any open response activities, the total number of minutes during the past 2 weeks is divided by 60 minutes, and then by 2, to determine the number of hours of physical activity per week. The minimum composite index is 0. A higher composite index indicates more physical activity.
Functional Dependence (Physical functioning) | Phase I at 1 month
  US Health Interview Survey - assesses engagement in physical activities in the prior two weeks. A composite index of physical activity is computed by summing the products of the number of minutes in each activity (9 are listed and there is an open response "other" option) and how many times in the past two weeks the engaged in the activity for the 9 activities and any open response activities, the total number of minutes during the past 2 weeks is divided by 60 minutes, and then by 2, to determine the number of hours of physical activity per week. The minimum composite index is 0. A higher composite index indicates more physical activity.
Functional Dependence (Physical functioning) | Phase I at 3 months
  US Health Interview Survey - assesses engagement in physical activities in the prior two weeks. A composite index of physical activity is computed by summing the products of the number of minutes in each activity (9 are listed and there is an open response "other" option) and how many times in the past two weeks the engaged in the activity for the 9 activities and any open response activities, the total number of minutes during the past 2 weeks is divided by 60 minutes, and then by 2, to determine the number of hours of physical activity per week. The minimum composite index is 0. A higher composite index indicates more physical activity.
Functional Dependence (Physical functioning) | Phase II at baseline
  US Health Interview Survey - assesses engagement in physical activities in the prior two weeks. A composite index of physical activity is computed by summing the products of the number of minutes in each activity (9 are listed and there is an open response "other" option) and how many times in the past two weeks the engaged in the activity for the 9 activities and any open response activities, the total number of minutes during the past 2 weeks is divided by 60 minutes, and then by 2, to determine the number of hours of physical activity per week. The minimum composite index is 0. A higher composite index indicates more physical activity.
Functional Dependence (Physical functioning) | Phase II at 3 months
  US Health Interview Survey - assesses engagement in physical activities in the prior two weeks. A composite index of physical activity is computed by summing the products of the number of minutes in each activity (9 are listed and there is an open response "other" option) and how many times in the past two weeks the engaged in the activity for the 9 activities and any open response activities, the total number of minutes during the past 2 weeks is divided by 60 minutes, and then by 2, to determine the number of hours of physical activity per week. The minimum composite index is 0. A higher composite index indicates more physical activity.
Functional Dependence (Physical functioning) | Phase II at 6 months
  US Health Interview Survey - assesses engagement in physical activities in the prior two weeks. A composite index of physical activity is computed by summing the products of the number of minutes in each activity (9 are listed and there is an open response "other" option) and how many times in the past two weeks the engaged in the activity for the 9 activities and any open response activities, the total number of minutes during the past 2 weeks is divided by 60 minutes, and then by 2, to determine the number of hours of physical activity per week. The minimum composite index is 0. A higher composite index indicates more physical activity.
Behavioral Activation Scale | Phase I at baseline.
  8 items based on Kanter et al., 2007 behavioral activation for depression scale. 1 item developed and added per researcher discretion. Responses range from 0 (meaning not at all) to 6 (meaning completely). Two items are reverse coded. Scores at each time point will be averaged.
Behavioral Activation Scale | Phase I at 1 month.
  8 items based on Kanter et al., 2007 behavioral activation for depression scale. 1 item developed and added per researcher discretion. Responses range from 0 (meaning not at all) to 6 (meaning completely). Two items are reverse coded. Scores at each time point will be averaged.
Behavioral Activation Scale | Phase I at 3 months.
  8 items based on Kanter et al., 2007 behavioral activation for depression scale. 1 item developed and added per researcher discretion. Responses range from 0 (meaning not at all) to 6 (meaning completely). Two items are reverse coded. Scores at each time point will be averaged.
Behavioral Activation Scale | Phase II at baseline.
  8 items based on Kanter et al., 2007 behavioral activation for depression scale. 1 item developed and added per researcher discretion. Responses range from 0 (meaning not at all) to 6 (meaning completely). Two items are reverse coded. Scores at each time point will be averaged.
Behavioral Activation Scale | Phase II at 3 months.
  8 items based on Kanter et al., 2007 behavioral activation for depression scale. 1 item developed and added per researcher discretion. Responses range from 0 (meaning not at all) to 6 (meaning completely). Two items are reverse coded. Scores at each time point will be averaged.
Behavioral Activation Scale | Phase II at 6 months.
  8 items based on Kanter et al., 2007 behavioral activation for depression scale. 1 item developed and added per researcher discretion. Responses range from 0 (meaning not at all) to 6 (meaning completely). Two items are reverse coded. Scores at each time point will be averaged.
Utilization of Unpaid Social Support Care Resources | Phase I at baseline.
  10-item yes or no checklist developed based on Kasper et al., 2015. 1 additional open-ended item is added to ask about other forms of unpaid social support. The total number of yes responses for each participant will be summed at each time point.
Utilization of Unpaid Social Support Care Resources | Phase I at one month.
  10-item yes or no checklist developed based on Kasper et al., 2015. 1 additional open-ended item is added to ask about other forms of unpaid social support. The total number of yes responses for each participant will be summed at each time point.
Utilization of Unpaid Social Support Care Resources | Phase I at three months.
  10-item yes or no checklist developed based on Kasper et al., 2015. 1 additional open-ended item is added to ask about other forms of unpaid social support. The total number of yes responses for each participant will be summed at each time point.
Utilization of Unpaid Social Support Care Resources | Phase II at baseline.
  10-item yes or no checklist developed based on Kasper et al., 2015. 1 additional open-ended item is added to ask about other forms of unpaid social support. The total number of yes responses for each participant will be summed at each time point.
Utilization of Unpaid Social Support Care Resources | Phase II at 3 months.
  10-item yes or no checklist developed based on Kasper et al., 2015. 1 additional open-ended item is added to ask about other forms of unpaid social support. The total number of yes responses for each participant will be summed at each time point.
Utilization of Unpaid Social Support Care Resources | Phase II at 6 months.
  10-item yes or no checklist developed based on Kasper et al., 2015. 1 additional open-ended item is added to ask about other forms of unpaid social support. The total number of yes responses for each participant will be summed at each time point.
Paid Service Use | Phase I at baseline.
  12-item measure assessing the utilization of paid community-based, residential, or other services. Response options include "I use this service," "I would like to use this service," and "I don't need to use this service." The number of services used will be summed at each time point for each participant.
Paid Service Use | Phase I at one month.
  12-item measure assessing the utilization of paid community-based, residential, or other services. Response options include "I use this service," "I would like to use this service," and "I don't need to use this service." The number of services used will be summed at each time point for each participant.
Paid Service Use | Phase I at three months.
  12-item measure assessing the utilization of paid community-based, residential, or other services. Response options include "I use this service," "I would like to use this service," and "I don't need to use this service." The number of services used will be summed at each time point for each participant.
Paid Service Use | Phase II at baseline.
  12-item measure assessing the utilization of paid community-based, residential, or other services. Response options include "I use this service," "I would like to use this service," and "I don't need to use this service." The number of services used will be summed at each time point for each participant.
Paid Service Use | Phase II at 3 months.
  12-item measure assessing the utilization of paid community-based, residential, or other services. Response options include "I use this service," "I would like to use this service," and "I don't need to use this service." The number of services used will be summed at each time point for each participant.
Paid Service Use | Phase II at 6 months.
  12-item measure assessing the utilization of paid community-based, residential, or other services. Response options include "I use this service," "I would like to use this service," and "I don't need to use this service." The number of services used will be summed at each time point for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Gaugler, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Study data and appropriate study materials/documentation will be deposited and made available through the National Archive of Computerized Data on Aging (NACDA), a NIA/NIH funded repository.
Access Criteria: Data and supporting documents/materials will be deposited in the NACDA repository.